CLINICAL TRIAL: NCT07111585
Title: Effect of Personalized Health Coaching Program in Patients With Frailty and Heart Failure
Brief Title: Personalized Health Coaching for Patients With HF
Acronym: Coach-FrailHF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gachon University Gil Medical Center (Other)
Responsible Party: Principal Investigator, Wook-Jin Chung, Professor, Gachon University Gil Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: WJC-IIT-1003
Record Dates: First submitted 2025-06-23; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-07

CONDITIONS: Heart Failure; Frailty; Health Coaching; Telenursing; Patient Monitoring; Randomized Controlled Trial
MeSH Terms: conditions — Heart Failure; Frailty | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized health coaching program (Experimental)
  Interventions: Other: Personalized health coaching program
- standard care (Other)
  Interventions: Other: standard care

INTERVENTIONS:
Other: Personalized health coaching program — Clinical: Pre-discharge education on HF management (e.g., symptoms, treatment, diet, medication, lifestyle) is provided with a booklet and website link. A digital scale is given. After discharge, 12-week phone coaching monitors medication adherence, weight, and sodium intake.
  Functional: Patients are referred to cardiac rehab for tailored exercise plans. Education on home exercise and oxygen monitoring is provided, with QR-linked videos. Coaching supports exercise adherence.
  Psycho-cognitive: Emotional support is based on the PERMA model. Patients with severe issues are referred to psychiatry. Post-discharge, coaching includes psychiatric appointment support and use of the 100-Day Diary for self-care and gratitude journaling.
  Social: Nurses foster trust and social reintegration. Referrals to community services are made as needed. Weekly calls ensure service connection and address unmet needs via social workers.
  Arms: Personalized health coaching program
Other: standard care — Participants in the control group will receive standard care, including guideline-directed medical therapy, based on the latest clinical guidelines currently provided to patients with HF at the hospital, as well as HF education. HF education will be provided using a booklet that includes information on HF (definition, causes, symptoms, diagnosis, treatment, medications, and self-management), an exercise poster, a symptom log, a symptom checklist, fall prevention tips, and a dietary guide. Additionally, nutritionist consultations on HF-related diets, cardiac rehabilitation exercises, and financial support available through the social work department, if necessary, will be provided.
  Arms: standard care

SUMMARY:
Frailty in heart failure (HF) patients contributes to poor outcomes, emphasizing the need for effective management. In many previous studies, frailty interventions have mainly targeted physical frailty or focused community-dwelling patients, neglecting the multidimensional needs of hospitalized individuals. As a frailty for HF patients need to include clinical, functional, cognitive, and social domains, nurses must assess it holistically and provide personalized support, especially during care transitions. This study aims to evaluate the effectiveness of a nurse-led, personalized health coaching program for hospitalized HF patients with frailty through a randomized controlled trial. This 12-week intervention program targets hospitalized HF patients with frailty. After screening frailty HF patients using validated tools such as Fried's phenotype (FP), Tilburg Frailty Indicator (TFI), participants will be randomly assigned to either an intervention or control group. The intervention group will receive personalized health services, including pre-discharge education and weekly telephone coaching, addressing clinical, functional, psycho-cognitive, and social frailty domains. Psychiatric support and community integration program will be provided as needed. The control group will receive standard care. Frailty, QoL, and clinical outcomes will be measured at baseline, 12 weeks, and 24 weeks. The primary outcomes will be improvements in frailty and QoL. Frailty will be measured both multidimensional and each of the four domains of frailty for HF patients. This study will clarify the role of multidimensional personalized interventions in addressing adverse outcomes related to frailty in patients with HF, thereby providing evidence of their necessity in its management.

DETAILED DESCRIPTION:
The prevalence of heart failure (HF) is increasing worldwide, and consistently in Korea, it has more than tripled between 2002 and 2020. As a result, the hospitalization rate due to HF has increased by 1.6 times, and the age-standardized mortality rate by more than fivefold. Despite the implementation of various treatment and management strategies, hospitalizations, unplanned visits and mortality related to HF continue to rise, underscoring the urgent need for multidimensional and personalized approaches to patient care. Particularly in Korea, the prevalence of HF begins to rise in an individual's 30s, and shows a significant increase after the age of 40s, with mortality rates gradually upward among middle-aged patients. Thus, there is the need to focus on health care among patients aged 40 and over.

One of the most common and critical issues observed in patients with HF is frailty. In HF, frailty is defined as a multidimensional, dynamic, and potentially reversible condition that, although age-related, is distinct from aging, that increases susceptibility to stressors and adverse outcomes. The overall prevalence of frailty among HF patients is estimated round 44.5%, although varying among measurement tools. Patients with frailty and HF exhibit a higher risk of cardiovascular death, HF-related hospitalization, all-cause death, and all-cause hospitalization as well as a lower quality of life (QoL). Although frailty is often age-related, it is not exclusive to the elderly, making frailty assessment essential for all patients with HF. Most existing frailty assessment tools emphasize only physical aspects and fail to capture the complexity of frailty in HF patients. Therefore, it is essential to plan and evaluate patients care using a multidimensional approach encompassing clinical, functional, cognitive-psychological, and social domains, as recommended by HF associations, which may help prevent or reduce adverse clinical outcomes.

According to the research results conducted so far, the evidence that multidimensional interventions more effectively improve frailty than single-domain interventions have been consisted, and a variety of healthcare professionals have delivered collaborative interventions to improve frailty. Among theses, nurse-led multidimensional interventions for community-dwelling older adults have shown improvements in frailty, physical function, nutritional status, QoL, social support, and mental health including reduced depression. In inpatient settings, nurses might play a key role in multidisciplinary teams as skilled health professional, educators, care coordinators, patient advocates, and liaisons. Therefore, HF nurses are able to plan and implement personalized interventions tailored to patients' individual needs in a central role.

The period from hospital admission to discharge is the most appropriate time to plan transition from hospital to home and a critical window for multidisciplinary intervention with HF patients. During hospitalization, above all else patients are at a high-risk stage of HF progress and frailty, and so early identification and fast management of HF progress are crucial. But most multidimensional interventions for frailty in HF have been conducted in community-based settings with no connection from the time of hospitalization. Hospital HF nurses can closely monitor patients' frailty status, coordinate with the care team, and plan for effective care transitions post-discharge. A structured transitional care strategy can help HF patients to maintain health care management and prevent readmissions at home.

Health coaching has emerged as an effective, goal-oriented, and patient-centered approach to support post-discharge self-care and behavior modification. After discharge interventions through phone calls, home visits, outpatient visit, or remote monitoring are essential components of HF management programs. A meta-analysis found that telecoaching has a significant impact on health outcomes, improving self-care and QoL in patients with HF. One study demonstrated that a 3-month personalized coaching program significantly reduced emergency visits and 6-month readmission rates, highlighting the importance of time in effecting behavioral change. Another study indicated that while younger patients prefer mobile or text-based interventions, older adults are more inclined to use telephone coaching in combination with paper-based health summaries. Thus, telephone coaching with paper manual book might be a particularly effective intervention for older, frail HF patients.

This study aims to present a protocol for evaluating the effects of a personalized telephone-based health coaching program on frailty, health-related QoL, and clinical outcomes among older patients hospitalized with heart failure. The findings are expected to contribute to the development of a practical, nurse-led inpatient intervention model that enhances the quality of HF patient care.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 40 years or older will be included in the study, as heart failure (HF)-related mortality and the prevalence of HF increase significantly from this age onward. Inclusion criteria requires a diagnosis of acute HF by a cardiologist and hospitalization based on the following criteria: presence of HF symptoms (e.g., breathlessness, fatigue, ankle swelling) and signs (e.g., elevated jugular venous pressure, pulmonary crackles, peripheral edema), evidence of pulmonary congestion or edema on chest X-ray, and elevated levels of BNP (≥100 pg/mL) or NT-proBNP (≥300 pg/mL). After initial screening for frailty using both the Tilburg Frailty Indicator (TFI) and Fried's Phenotype (FP), participants will be enrolled if they are classified as frail, able to cooperate with functional assessments, and willing to provide written informed consent with a clear understanding of the study's purpose and procedures.

Exclusion Criteria:

* The exclusion criteria were as follows: current enrollment in other programs or planning to participate in similar programs during the intervention period; residing outside Korea and not understanding Korean; diagnosis of dementia with the Global Deterioration Scale stage of 5 or greater; inability to comprehend the study purpose and content.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-07-03 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Clinical Frailty Scale (CFS) | Baseline assessment, Mid assessment (6 week), Post assessment (12 week), Final assessment (24 week)
  The CFS measures frailty using a quick assessment through brief descriptions and illustrations. The total score ranges from 1 to 9, with a score of ≥4 indicating frailty.
Kansas City Cardiomyopathy Questionnaire clinical summary score (KCCQ-CSS) | Baseline assessment, Mid assessment (6 week), Post assessment (12 week), Final assessment (24 week)
  The Clinical Summary Score (CSS) is calculated as the mean of the Physical Limitation Score and the Total Symptom Score from the KCCQ. The KCCQ CSS ranges from 0 to 100, where higher scores indicate better health status.

SECONDARY OUTCOMES:
Tilburg Frailty Indicator (TFI) | Baseline assessment, Post assessment (12 week), Final assessment (24 week)
  The TFI was developed based on an integral conceptual model of frailty that categorizes it into 3 dimensions: physical (8 items), psychological (4 items), and social (3 items). The frailty score (maximum, 15) is determined by summing the scores of the 3 frailty domains. Frailty is identified as a score ≥5.
Frailty phenotype (FP) | Baseline assessment, Post assessment (12 week), Final assessment (24 week)
  The FP included the following 5 criteria: loss of muscular strength (grip strength), reduced gait speed, weight loss, exhaustion, and reduced physical activity. A pre-frail state is identified when a patient meets 1 or 2 of these criteria, whereas a frail state is identified when a patient meets more than 2 criteria. Specifically, grip strength was measured using a Jamar hydraulic dynamometer, the gold standard for grip strength assessment.
Frailty Idex-Laboratory (FI-laboratory) | Baseline assessment, Post assessment (12 week), Final assessment (24 week)
  The FI-Laboratory measures frailty based on routine physical assessments and blood tests based on the accumulation of deficits. Each item was scored between 0 and 1, with 0 and 1 indicating ideal health and a theoretical state of complete frailty, respectively. The total score was calculated by dividing the total number of items assessed by the sum of the deficit item scores, with higher scores reflecting increased frailty
Mini-Cog | Baseline assessment, Post assessment (12 week), Final assessment (24 week)
  The Mini-Cog, which is used to screen for cognitive issues, comprises 3 components-3-word registration, clock drawing, and 3-word recall-with a maximum score of 5. One point was assigned for each accurately recalled word (total of 3 points), whereas 2 points were assigned for accurately drawing the clock. A score of ≤2 indicates the presence of cognitive problems
Patient Health Questionnaire-9 (PHQ-9) | Baseline assessment, Post assessment (12 week), Final assessment (24 week)
  The PHQ-9 measures depression and comprises 9 items rated from 0 (not at all) to 3 (nearly every day). The maximum total score is 27, with scores of 10-19 and 20-27 indicating moderate and severe depression, respectively
Makizako Social Frailty Index | Baseline assessment, Post assessment (12 week), Final assessment (24 week)
  The Makizako Social Frailty Index measures social frailty and comprises 5 items, with 2 or more positive responses to questions indicating social frailty.
Heart Failure Frailty Scale (HFFS) | Baseline assessment, Post assessment (12 week), Final assessment (24 week)
  The HFFS is a multidimensional frailty assessment instrument that was developed specifically for patients with HF4) and comprises 4 domains. As of now, no validated cut-off score has been universally established to classify frailty status.
Kansas City Cardiomyopathy Questionnaire | Baseline assessment, Post assessment (12 week), Final assessment (24 week)
  The KCCQ comprises 23 items that quantify 7 domains-physical limitations (6 items), symptom stability (1 item), symptom frequency (4 items), symptom burden (3 items), self-efficacy (2 items), QoL (3 items), and social limitations (4 items)-of health status in patients with HF. Scores range from 0 to 100, with higher scores indicating better health status and quality of life.
Worsening Heart Failure events | Baseline assessment, Post assessment (12 week), Final assessment (24 week)
  hospitalizations, emergency room visits, and unscheduled visits to outpatients' clinics
Change in NT-proBNP Level from Baseline | Baseline assessment, Post assessment (12 week), Final assessment (24 week)
Change in New York Heart Association Functional Class from Baseline | Baseline assessment, Post assessment (12 week), Final assessment (24 week)
  Assessed by the New York Heart Association (NYHA) Functional Classification, ranging from Class I to Class IV, with higher classes indicating worse functional status.
6-minute walk distance | Baseline assessment, Post assessment (12 week), Final assessment (24 week)
changes in muscle mass measured by impedance | Baseline assessment, Post assessment (12 week), Final assessment (24 week)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiovascular Medicine, Gachon University, Gil Medical Center, Incheon,, Incheon, South Korea

IPD SHARING:
Plan to Share IPD: No